CLINICAL TRIAL: NCT00812396
Title: A Randomized, Single-Blind, Placebo-Controlled, Fixed-Sequence, Single-Dose, Parallel Design Study to Utilize Comparative Proteomics to Identify Early Biomarkers of Muscle Anabolism
Brief Title: Biomarkers of Muscle Anabolism (MK-0000-082)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0000-082; 2008_602
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Muscle Anabolism
Keywords: Biomarkers of muscle anabolism
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Low dose testosterone
  Interventions: Drug: Comparator: low dose testosterone
- 2 (Active Comparator): High dose testosterone
  Interventions: Drug: Comparator: high dose testosterone
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: Comparator: low dose testosterone — Subjects will receive two muscle biopsies, the first at baseline, and the second a week after a single intramuscular dose of 200 mg (0.8 mL) testosterone.
  Arms: 1
Drug: Comparator: high dose testosterone — Subjects will receive two muscle biopsies, the first at baseline, and the second a week after a single intramuscular dose of 600 mg (2.4 mL) testosterone.
  Arms: 2
Drug: Comparator: placebo — Subjects will receive two muscle biopsies, the first at baseline, and the second a week after a single intramuscular dose of 0.8 mL placebo saline solution.
  Arms: 3

SUMMARY:
This study will evaluate the ability of comparative proteomics to identify early biomarkers of muscle anabolism.

ELIGIBILITY:
Inclusion Criteria:

* subject is a healthy male between 18 and 40 years old
* subject's weight is stable over the past 3 months
* subject agrees to refrain from consuming alcohol during study
* subject agrees to consume no caffeine while in the CRU
* subject agrees to follow meat-free diet
* subject is willing to avoid strenuous activity
* subject has been a nonsmoker for at least 6 months

Exclusion Criteria:

* subject is a regular user of illicit drugs
* subject has taken androgenic steroids in the past 12 months
* subject has participated in sports events, resistance training, or moderate to heavy endurance training in the past month
* subject has prostate cancer
* subject has HIV and/or hepatitis B or C

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
comparative proteomics on proteins present in the vastus lateralis or plasma | 1 week

SECONDARY OUTCOMES:
mRNA or miRNA expression in the vastus lateralis or in peripheral blood | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Chen F, Lam R, Shaywitz D, Hendrickson RC, Opiteck GJ, Wishengrad D, Liaw A, Song Q, Stewart AJ, Cummings CE, Beals C, Yarasheski KE, Reicin A, Ruddy M, Hu X, Yates NA, Menetski J, Herman GA. Evaluation of early biomarkers of muscle anabolic response to testosterone. J Cachexia Sarcopenia Muscle. 2011 Mar;2(1):45-56. doi: 10.1007/s13539-011-0021-y. Epub 2011 Feb 26. PMID 21475673